CLINICAL TRIAL: NCT05824169
Title: A Multi-center, Open Label, Single-arm, Dose Ascending Clinical Trial for Evaluation of Safety and Efficacy of Gene Therapy Drug GC101 in the Treatment of Spinal Muscular Atrophy (SMA) Type 1 Patients
Brief Title: Evaluation of Safety and Efficacy of Gene Therapy Drug in the Treatment of Spinal Muscular Atrophy (SMA) Type 1 Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GeneCradle Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JLJY-GC101-SMA-001
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Spinal Muscular Atrophy
Keywords: Type 1
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dosage group (Experimental): 2.4x10^14 vg/person of GC101 delivered one-time intrathecally (n=3)
  Interventions: Genetic: GC101
- High dosage group (Experimental): 4.8x10^14 vg/person of GC101 delivered one-time intrathecally (n=3)
  Interventions: Genetic: GC101

INTERVENTIONS:
Genetic: GC101 — Self-complementary AAV9 carrying a codon-optimized SMN coding sequence(coSMN1) driven by CMV enhancer and chicken β-actin promoter

SUMMARY:
The study will evaluate safety and efficacy of intrathecal delivery of GC101 gene therapy drug as a treatment of spinal muscular atrophy Type 1 (SMA 1) patients.

DETAILED DESCRIPTION:
The purpose of this trial is to evaluate safety and efficacy of gene therapy drug GC101 in SMA 1 patients. Open-label, dose-escalation clinical trial of GC101 will be conducted in multiple centers in China.

GC101 will be administrated intrathecally. Short-term safety will be evaluated in 52 weeks and enter long-term follow-up study of 5 years at will. Patients will be tested at baseline and followed up on various time points.

The primary analysis for efficacy will be assessed when all patients reach 18 months of age on the motor milestone of sit unassisted for at least 10 seconds.

ELIGIBILITY:
Inclusion Criteria:

* Six months of age and younger on day of vector infusion with Type 1 SAM as defined by the following features:

  * Diagnosis of SMA based on gene mutation analysis with bi-allelic SMN1 mutations (deletion or point mutations) and 2 copies of SMN2;
  * Onset of disease before 6 months of age
* The patient's legal guardian(s) must be able to understand the purpose and risks of the study and voluntarily provide signed and dated informed consent prior to any study-related procedures being performed.

Exclusion Criteria:

* Patient who has participated in a previous gene therapy research trials;
* Patient who has received Nusinersen and Risdiplam treatment;
* Patient who has AAV9 neutralizing antibody titer ≥1:200;
* Patient who requires non-invasive ventilatory support averaging≥16 hours/day;
* Patient with a point mutation in SMN2 (c.859G>C);
* Patient who requires non-invasive ventilatory support averaging≥16 hours/day at screening;
* Patient who use invasive ventilatory support or pulse oximetry < 95% saturation while awake and calm at screening;
* Patient who is positive for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, hepatitis C antibody, or treponema pallidum antibody;
* Abnormal laboratory values considered clinically significant, including gamma-glutamyl transferase(GGT), Aspartate aminotransferase (AST), alanine aminotransferase (ALT), bilirubin > 3x upper limit of normal (ULN), Hemoglobin (Hgb)< 110 or >150 g/L, platelet <183x10^9/L or 614x10^9/L;
* Class IV patient based on Modified Ross Heart Failure Classification for Children;
* Patient with a history of glucocorticoid allergy;
* Contraindication that would interfere with the lumbar puncture procedures;
* Presence of an untreated active infection requiring systemic antiviral therapy at any time during the screening period;
* Vaccination less than 2 weeks before infusion of vector;
* Patient who has any concurrent clinically significant major disease or any other condition that, in the opinion of the Investigator, makes the subject unsuitable for participation in the study.

Note: Other protocol defined inclusion/exclusion criteria may apply.

Ages: 0 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2023-02-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | when patient reaches 18 months of age
  Frequency of treatment-related adverse events (AEs), serious adverse events (SAEs), and changes from baseline in relevant clinical laboratory tests
Proportion of patients treated with GC101 who achieve motor milestone of sit unassisted for at least 10 seconds at 18 months of age | when patient reaches 18 months of age

SECONDARY OUTCOMES:
Ability to thrive | when patient reaches 18 months of age
  Ability to thrive is defined as the following at 18 months of age: does not receive nutrition through mechanical support or other non-oral method; maintains weight
Changes from baseline Children's hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP-INTEND) score | when patient reaches 18 months of age
  CHOP INTEND score ranges from 0 to 64 with higher scores indicating higher motor function
Proportion of event-free survival patients | when patient reaches 14 months of age

OTHER OUTCOMES:
Proportion of patients who achieve the World Health Organization (WHO) Multicenter Growth Reference Study (MGRS) motor milestones | when patient reaches 18 months of age
  WHO MGRS gross motor milestones and performance criteria included sitting without support for at least 10 seconds, Hands-and-knees crawling at least three in a row, standing with assistance for at least 10 seconds, walking with assistance at least five steps, standing alone for at least 10 seconds, and walking alone.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Peking University， First Hospital, Department of Pediatrics, Beijing
  - Bayi Children's Hospital, Seventh Medical Center, PLA general hospital, Beijing
  - Shengjing Hospital of China Medical University, Shenyang
  - Children's Hospital of Soochow University, Suzhou

IPD SHARING:
Plan to Share IPD: No